CLINICAL TRIAL: NCT04194853
Title: Effects of Electromyographic Biofeedback on Performance of Vastus Medialis Oblique Muscle in Knee Osteoarthritis
Brief Title: Electromyographic Biofeedback on Performance of Vastus Medialis Oblique Muscle in Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RiphahIU Huma Khan
Record Dates: First submitted 2019-11-20; First posted 2019-12-11 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: There will be two treatment groups of participants, Experimental group will receive Isometric exercises with EMGBF( Electromyographic Biofeedback ) and control group receive exercises without EMGBF.
Who Masked: Participant
Masking Description: There will be two treatment groups of participants, Experimental group will receive Isometric exercises with EMGBF( Electromyographic Biofeedback ) and control group receive exercises without EMGBF.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EMG Biofeedback assisted Quadriceps exercises. (Experimental): Hot Pack will be applied before session for general relaxation for 10 minutes. Knee isometric exercises will be performed via an EMG Biofeedback device; patients in the EMG BF group will receive visual and auditory feedback.Knee isometrics will be performed with 5 seconds hold. Then, the muscle will be relaxed for 10 seconds and the cycle repeated for a total of 15 minutes. (20 reps, 3 sets) Session will be performed thrice a week for six weeks.
  Interventions: Device: Electromyographic Biofeedback
- Quadriceps exercises without EMG Biofeedback (Active Comparator): Hot Pack will be applied before session for general relaxation 10 minutes. In the control group, the active electrode will not be connected, so subjects will not receive any feedback from the device. Knee isometrics perform with 5 seconds hold. Then, the muscle will be relaxed for 10 seconds and the cycle repeated for a total of 15 minutes. (20 reps, 3 sets)Session will be performed thrice a week for six weeks.
  Interventions: Other: Quadriceps Isometric exercises

INTERVENTIONS:
Device: Electromyographic Biofeedback — Surface EMG biofeedback is an adjunct therapy to standard exercise regime for increasing muscle strength .Electromyographic (EMG) biofeedback is a specific form of biofeedback. The biofeedback device records muscle activity through the application of electrodes superficially or subcutaneously when targeting specific muscles
  Arms: EMG Biofeedback assisted Quadriceps exercises.
Other: Quadriceps Isometric exercises — In supine lying or sitting, Patient is asked to press down knee while contracting Quadriceps muscles.
  Arms: Quadriceps exercises without EMG Biofeedback

SUMMARY:
This study intends to determine the Effects of Electromyographic biofeedback on performance of vastus medialis oblique muscle in knee osteoarthritis.

DETAILED DESCRIPTION:
This is a single blinded randomized controlled trial, will be conducted at Railway General Hospital.Rawalpindi.

(EMG) biofeedback as an adjunct therapy to standard exercise regime for increasing muscle strength ,this study is planned to determine the effects of electromyographic biofeedback on performance and thickness of vastus medialis oblique muscle, knee pain and on lower extremity function in patients with Knee Osteoarthritis. The sample size was calculated to be n=34 through Open Epi tool version 3, with 95 % confidence interval (CI), and power 80%.

After the completion of therapeutic protocols, the participants will be assessed with the help of Numeric Pain Rating Scale (NPRS), WOMAC, Lequesne questionnaire , 1 Repetition maximum( RM) and with MSK ultrasound

ELIGIBILITY:
Inclusion Criteria:

* Age : In between 45 - 65years
* Both Genders
* Subjects with a definite diagnosis of knee OA according to the guidelines of the American College of Rheumatology with at least 6 months of knee pain.
* Grade 1 or 2 joint cartilage degradation based on the Kellgren-Lawrence classification
* Body mass index (BMI) of <35 kg/m2

Exclusion Criteria:

* Subjects who had undergone physical therapy or intraarticular injection in the past 3 months
* Patients who had taken oral corticosteroids in the past 4 weeks
* Patients with a history of surgical interventions on their knees
* Subjects with a history of radiculopathy, or those with a history of systemic diseases, such as rheumatoid arthritis

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-01-03 (Actual); Study Completion 2020-01-08 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | Post 6 Weeks
  Changes from the baseline, Numeric Pain Rating Scale (NPRS) is used to assess pain. It scores ranges from 0-10, 0 means No pain and 10 means Severe pain. Patient will be asked to verbally report the pain score.
1 Repetition Maximum | Post 6th week
  Changes from the baseline, 1 RM Is used to assess maximum muscle strength. Patient is asked to extend knee against maximum resistance once.
Vastus medialis Oblique(VMO) Thickness | Post 6th week
  Changes from the Baseline, Musculoskeletal ultrasound will be used to measure maximum thickness of VMO muscle. Assessment will be done by a Consultant radiologist using a 7-12 MHz probe

SECONDARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | Post 6 weeks
  Changes from the baseline, WOMAC is used to assess the functional status. The questionnaire includes five questions about pain severity (0-20), two items on joint stiffness (0-8), and 17 questions on functional limitations of the patient (0-68). Each item is scored on a scale of 0-4, and the greater the score, the worse the pain and function. The total score of the subjects from this index was reported from a total of 96.

CONTACTS AND LOCATIONS:
Overall Officials: Huma Riaz, PHD*, Principal Investigator — Riphah International University
Locations (1):
- Pakistan Railway hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Raeissadat SA, Rayegani SM, Sedighipour L, Bossaghzade Z, Abdollahzadeh MH, Nikray R, Mollayi F. The efficacy of electromyographic biofeedback on pain, function, and maximal thickness of vastus medialis oblique muscle in patients with knee osteoarthritis: a randomized clinical trial. J Pain Res. 2018 Nov 8;11:2781-2789. doi: 10.2147/JPR.S169613. eCollection 2018. PMID 30519081
- [Background] Choi YL, Kim BK, Hwang YP, Moon OK, Choi WS. Effects of isometric exercise using biofeedback on maximum voluntary isometric contraction, pain, and muscle thickness in patients with knee osteoarthritis. J Phys Ther Sci. 2015 Jan;27(1):149-53. doi: 10.1589/jpts.27.149. Epub 2015 Jan 9. PMID 25642061
- [Background] Eid MA, Aly SM, El-Shamy SM. Effect of Electromyographic Biofeedback Training on Pain, Quadriceps Muscle Strength, and Functional Ability in Juvenile Rheumatoid Arthritis. Am J Phys Med Rehabil. 2016 Dec;95(12):921-930. doi: 10.1097/PHM.0000000000000524. PMID 27149595
- [Background] Florencio LL, Martins J, da Silva MRB, da Silva JR, Bellizzi GL, Bevilaqua-Grossi D. Knee and hip strength measurements obtained by a hand-held dynamometer stabilized by a belt and an examiner demonstrate parallel reliability but not agreement. Phys Ther Sport. 2019 Jul;38:115-122. doi: 10.1016/j.ptsp.2019.04.011. Epub 2019 Apr 25. PMID 31091492